CLINICAL TRIAL: NCT03213717
Title: Effect of Body Weight Loading on Urinary Electrolyte Excretion
Acronym: EBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EBU
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Edema
Keywords: Obesity; Loading; Edema; Urine
MeSH Terms: conditions — Obesity; Edema | interventions — Standing Position; Sitting Position

STUDY DESIGN:
Intervention Model Description: The study is executed with all 15 study subjects over three study days with one week between each study day. In order to decrease the variation of the measurement values and increase the power of the study we will use a cross-over study design. The study subjects will on one of the days wear a weight vest with 10 % of body weight in the standing position, on one of the days the same study subject will wear a weight vest with 1 % of body weight in the standing position and on one of the days the same study subject will wear a weight vest with 1 % of body weight in the sitting position.
  Hence, three procedures are included in the study. Each of the procedure corresponds to a separate day.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: We will recruit healthy individuals who work at or close to the Institution of Neuroscience and Physiology at the Sahlgrenska Academy. We will ask healthy people who do not know the hypothesis of the study. Each study subject will be given a randomized code to use for the study. Only the study subject and the investigator will be able to connect each study subject with their randomized code. This will only be used under special circumstances, for example, if a study subject requests removal of his or her study data.
  As this study uses a cross-over design each subject will then be its own matched control.
  Subject eligibility will be established before enrolment and randomization. Subjects will be randomized strictly sequentially, as subjects are eligible for randomization. If a subject discontinues from the study, the subject number will not be reused, and the subject will not be allowed to re-enter the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Procedure 1 (Experimental): Wearing a weight vest with 10 % of body weight standing for seven hours. The study subject is allowed to sit for 10 minutes each hour. The reason for this is because it has been considered that the effect may be transmitted by weight loading of the lower extremities.
  Interventions: Other: Heavy Casall HIT weight vest; Behavioral: Standing; Dietary Supplement: Water load
- Procedure 2 (Active Comparator): Wearing a weight vest with 1 % of body weight standing for seven hours. The study subject is allowed to sit for 10 minutes each hour.
  Interventions: Behavioral: Standing; Dietary Supplement: Water load; Other: Light Casall HIT weight vest
- Procedure 3 (Active Comparator): Wearing a weight vest with 1 % of body weight sitting for seven hours. This is a control group without loading of the lower extremities. This is also the normal working position for many sedentary jobs (e.g. office workers) and why this is of special interest for further investigation. There is a large body of investigative literature showing the negative health consequences of the sitting working position.
  Interventions: Dietary Supplement: Water load; Behavioral: Sitting; Other: Light Casall HIT weight vest

INTERVENTIONS:
Other: Heavy Casall HIT weight vest — A weight west with a weight of 10 % compared to the study subject
  Arms: Procedure 1
Behavioral: Standing — Study subjects will be standing for at least 50 minutes every hour
  Arms: Procedure 1; Procedure 2
Dietary Supplement: Water load — Study subjects will drink 5 ml per kg body weight at the start of experiment and continue drinking the same volume as excreted by the kidneys during the experiment
Behavioral: Sitting — Study subjects will be sitting for at least 50 minutes of every hour
  Arms: Procedure 3
Other: Light Casall HIT weight vest — A weight west with a weight of 1 % compared to the study subject
  Arms: Procedure 2; Procedure 3

SUMMARY:
Title: Effect of body weight loading on urinary electrolyte excretion

Swedish Title: Effekt av belastning på utsöndring av elektrolyter

Study period: Q2-Q3 2017

Study site: The study will be performed at the Institution for Neurology and Physiology, Sahlgrenska Academy, University of Gothenburg. Principal Investigator is John-Olov Jansson, MD, PhD, Professor at Institute of Neuroscience and Physiology, University of Gothenburg

Background and study design: Weight reduction can be obtained by decreased appetite or increased metabolism. However, acute weight loss can also be obtained by loss of fluids - for example by increased urinary loss of fluid and salts, so called elctrolytes. Preliminary results from a laboratory lesson for the Master of Science in Medicine program at University of Gothenburg suggest that carrying a 10 kg weight vest could increase urinary excretion of Na+, K+ and Cl-. The purpose of this study is to investigate this further in a more controlled research setting. If confirmed, the results could potentially contribute to the development of potent diuretics or obesity medicines.

The study will include 15 healthy volunteers and consist of three study days with about one week between each study day. The study subjects will go through a different study procedure each study day, and a randomized cross-over study design will be used to determine which procedure each day.

Procedure 1: Wearing a weight vest with 10 % of body weight standing for seven hours. The study subject is allowed to sit for 10 minutes each hour. The reason for this is that it has been considered that the effect may be transmitted by weight loading of the lower extremities.

Procedure 2: Wearing a weight vest with 1 % of body weight standing for seven hours, as a control for procedure 1, with lower loading. The study subject is allowed to sit for 10 minutes each hour.

Procedure 3: Wearing a weight vest with 1 % of body weight sitting for seven hours. This is a procedure with even less loading of the lower extremities than during procedure 2.

Urine- and blood samples, as well as heart rate and blood pressure measurements, will be collected during the study days and analyzed in order to address the primary and secondary objectives of the study.

DETAILED DESCRIPTION:
1. INTRODUCTION

   1.1. Background

   Weight reduction can be obtained by decreased appetite or increased metabolism. However, acute weight loss can also be obtained by loss of fluids - for example, urinary loss. The last of these effects was investigated during 2016.

   The medical education at The Sahlgrenska Academy in Gothenburg offers in its third semester a student lab called "Vattenbalans" [=Water balance]. The purpose of this lab is to study fluid loss by the kidneys. In total more than 120 students participate, although the urine flow rate is only measured on approximately 50 students each semester. The rest of the students function as secretaries. The lab protocol can be found in "Komplett-laborationskompendium-T2-T3-uppdaterat-150318" pp. 123-134.

   In summary a total of 50 students wore a weight west. Half of the students wore a 10 kg weight vest and half of the students wore a 1 kg weight vest. The study lasted for four hours. The students were only allowed to sit a maximum of 10 minutes during each hour. No significant difference was observed in urine flow rate. Surprisingly however, the investigators found that the students who wore a 10 kg weight vest excreted more electrolytes than those wearing a 1 kg weight vest. In the group free from treatment (see below) only consisted of 13 subjects and the investigators were therefore not able to obtain significant results (p=0,088). The investigators believe that with a larger study population and better matched controls the investigators will reach significant results.

   It shall be noted that these results were obtained during a student lab with a fixed protocol. In addition to wearing a weight vest the students also received one of the following treatments: one liter of water orally, one liter of water orally and oral administration of a vasopressin analogue called Minirin© (desmopressin, 60 µg), a loop diuretic called Furix© (furosemide, 40 mg) or one liter water orally and eight tablets of Resorb© which is a rehydration therapy. The multiple treatments and the fixed protocol are confounders and support the repetition of these experiments with a more suitable design.

   1.2. Rationale for conducting this study

   The medical relevance of these experimental results is still unclear because of the short duration of four hours. With more experimental support, it is possible that this strategy could be used to create potent diuretics. It is also possible that long-term body weight loading could decrease body weight in a different way, especially by decreasing fat mass. This mechanism could therefore be used to create potent drugs for obesity.

   1.3. Risk/Benefit evaluation

   In general this is a study with few risks. The weight vests used in this experiment are in daily use by thousands of people during exercise . During the experiment with medical students only one of the students experienced an adverse event. This student experienced mild dizziness which subsided within a few minutes after removing the weight vest and sitting down. To further minimize the risks in our future study the investigatorshave decided to include only healthy research subjects consuming no medications. The investigators will also have medically trained personnel available during the study and perform it in close vicinity to the Sahlgrenska University Hospital.

   Blood sampling can be experienced as somewhat uncomfortable by a few individuals. However it is generally free from complications. In some subjects, there may be small local bruising or inflammation.

   In summary the investigators believe the risks to be very low compared to the potential of exploring a new physiological mechanism with potentially important applications such as new diuretics or anti-obesity medicine.
2. STUDY DESIGN AND PROCEDURES

The study is executed with all 15 study subjects over three study days with one week between each study day. In order to decrease the variation of the measurement values and increase the power of the study cross-over study design will be used. The study subjects will on one of the days wear a weight vest with 10 % of body weight in the standing position, on one of the days the same study subject will wear a weight vest with 1 % of body weight in the standing position and on one of the days the same study subject will wear a weight vest with 1 % of body weight in the sitting position.

Hence, three procedures are included in the study. Each of the procedure corresponds to a separate day.

Procedure 1: Wearing a weight vest with 10 % of body weight standing for seven hours. The study subject is allowed to sit for 10 minutes each hour. The reason for this is because it has been considered that the effect may be transmitted by weight loading of the lower extremities.

Procedure 2: Wearing a weight vest with 1 % of body weight standing for seven hours. The study subject is allowed to sit for 10 minutes each hour.

Procedure 3: Wearing a weight vest with 1 % of body weight sitting for seven hours. This is a control group without loading of the lower extremities. This is also the normal working position for many sedentary jobs (e.g. office workers) and why this is of special interest for further investigation. There is a large body of investigative literature showing the negative health consequences of the sitting working position.

Blood drawing will be performed with a peripheral venous catheter of the smallest size. Furthermore there will be several steps each day which will be uniform for each of the procedures.

Time point 1 (0 h): "Oral water load"

The catheter will be placed by an experienced nurse from Gothia Forum and is removed seven hours later when the procedure day is finished. Study proceedings and record keeping will be told to the research subject before the experiment officially starts.

Just before the experiment starts the study subject will drink 5 ml of water per kg body weight. For example, if the study subject weighs 70 kg (no weight vest), he or she will drink 350 ml of water.

To maintain a normal hydration level and urine production the study subject will continue to replace with fluids during the experiment. The volume of fluids that will be replaced will be equal to the amount of lost urine volume. If for example the study subject loses 100 ml urine he or she will drink of 100 ml water before continuing the experiment. By this method a urine production of approximately 200 ml per hour is maintained which is more than enough to perform all the required urine measurements.

This approach mimics physiological conditions wherein urinary losses are matched by water intake. It will avoid water intake in excess of replacement amounts which, in some circumstances, is viewed as treatment.

It is then decided by dice throw if a study subject will start with procedure 1, 2 or 3. When two of the procedure groups are full, with five individuals in each of them, the rest is transferred to the last procedure group. Rotation between the procedures occurs in random. Each study subject will have one week between performing each procedure.

The study subjects will empty their urine bladder just before the study starts. The study subjects start with five minutes separation to avoid congestioin to the toilets. The study starts when a study subject put on a weight vest.

Time Point 2 (0-7 h): Measurements and blood drawing

This time period consists of the part from when the study subject puts on the weight vest until the he or she takes it off.

The study subject shall each hour collect his or her urine volume in a specially designated measurement cup. The Urine Volume is noted. 10 ml of the urine are then used to measure the electrolyte concentration. Another 10 ml of urine is saved for further analyses at the Sahlgrenska University central lab. These analyses are routine but samples may be stored for a few days before the measurement takes place. This depends on when the central lab can accept our samples and on their specific working load. Sample storage and handling will be performed according to the central lab recommendations. The samples will at maximum be frozen down once at a temperature of -80°C.

When the urine measurements are complete the study subject will have five minutes to relax before measuring his or her heart rate and blood pressure. Heart rate and blood pressure are both measured standing and sitting with digital blood pressure monitors for quick and reliable values.

Blood will be drawn four times. The samples will be analyzed as soon as possible after each procedure day. Some analyses will be at the Sahlgrenska Academy directly, others will be delivered to Sahlgrenska University central lab (please see section 6.1 for details). These analyses are routine but samples may be stored for a few days before the measurement takes place. This depends on when the central lab can accept our samples and on their specific working load. Sample storage and handling will be performed according to the central labs recommendations.

Time point 3 (7 h -): The experiment is finished

Weight vest and peripheral venous catheter are removed. A procedure protocol is handed in from the study subject to the investigator who confirms its completeness. . The procedure protocol is either handed in digitally by uploading an excel file or handed in printed out.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects must fulfil the following criteria:

1. Healthy volunteers
2. Signed informed consent
3. Willingness to comply with study restrictions of not using alcohol, coffee etc during the hours specified below prior to each study day

Exclusion Criteria:

Subjects must not enter the study if any of the following are present:

1. Chronic disease requiring continuous medication or harden the participation in the study as judged by the investigator
2. High blood pressure (>140/90 mm Hg)
3. Chronic pain such as pain that is constant and impairs quality of life
4. Consumption of medications during the last 7 days prior the study day, not including contraceptives
5. Consumption of nature medicine or supplements that results in a increased intake of a specific compound that isn't a nutrient during the last 7 days prior the study day
6. Smoking, snuff use or intake of drugs during the last 7 days prior the study day
7. Intake of alcohol during the last 24 hours prior the study day
8. Intake of coffee and tea during the last 12 hours prior the study day
9. Strenuous physical activity before the study during the last 6 hours prior the study day
10. Pregnancy: Females of childbearing potential must confirm to use reliable contraception and not suspect to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Sodium concentration | 7 hours from start
  In urine

SECONDARY OUTCOMES:
Urine Volume | 7 hours from start
  ml
Potassium concentration | 7 hours from start
  in urine
Chloride concentration | 7 hours from start
  in urine
Calcium concentration | 7 hours from start
  in urine
Creatinine | 7 hours from start
  in urine
pH | 7 hours from start
  in urine
Sodium | 6.5 hours from start
  in serum
Potassium | 6.5 hours from start
  in serum
Chloride | 6.5 hours from start
  in serum
Creatinine | 6.5 hours from start
  in serum
Lipocalin2 | 6.5 hours from start
  in serum
Osteocalcin | 6.5 hours from start
  in serum
FGF23 | 6.5 hours from start
  in serum
Sclerostin | 6.5 hours from start
  in serum
Glucose | 6.5 hours from start
  in whole blood
Blood pressure | 7 hours from start
  Systolic and Diastolic (mmHg)
Heart Rate | 7 hours from start
  bpm

CONTACTS AND LOCATIONS:
Overall Officials: John-Olov Jansson, Principal Investigator — Univeristy of Gothenburg
Locations (1):
- University of Gothenburg, Gothenburg, Box 100, Sweden

IPD SHARING:
Plan to Share IPD: No